CLINICAL TRIAL: NCT05469347
Title: PCSK9 and Lipid Metabolism in Sepsis (PALMS) : a Two-center, Phase 1b Randomized, Placebo-controlled, Double-blind, Clinical Trial of Alirocumab in Patients with Sepsis
Brief Title: Alirocumab in Patients with Sepsis
Acronym: PALMS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonathan Sevransky (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Jonathan Sevransky, Professor, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00004119
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Sepsis
Keywords: Sepsis; Septic shock; Respiratory failure; Vasopressors
MeSH Terms: conditions — Sepsis; Shock, Septic; Respiratory Insufficiency | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alirocumab (Experimental): Critically ill participants with sepsis leading to cardiovascular and/or respiratory failure who are randomized to receive alirocumab.
  Interventions: Drug: Alirocumab
- Placebo (Placebo Comparator): Critically ill participants with sepsis leading to cardiovascular and/or respiratory failure who are randomized to receive a placebo to match alirocumab.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alirocumab — A 600 mg dose of alirocumab (which is equivalent to 8mg/kg for a 75kg patient) will be administered once via IV over an approximately 30 ± 10 minute infusion using an infusion pump.
  Other Names: Praluent
  Arms: Alirocumab
Drug: Placebo — A placebo to match a 600 mg dose of alirocumab will be administered once via IV over an approximately 30 ± 10 minute infusion using an infusion pump.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the drug alirocumab, which may lower cholesterol, can reduce the amount of inflammation caused by an infection that has caused either low blood pressure or difficulty breathing. Participants will be randomized to receive a single IV infusion of alirocumab or a placebo.

DETAILED DESCRIPTION:
Sepsis is an inflammatory syndrome with life threatening organ dysfunction resulting from a dysregulated host response to infection. The global burden is estimated to exceed 15 million cases annually. In the United States, the incidence is increasing and currently there are more 1,750,000 cases each year, with more than half requiring intensive care unit (ICU) admission. Further, sepsis cases account for 30%- 50% of all hospital deaths, making it the third leading cause of death in the United States, and is the most expensive reason for hospitalization with annual expenditures exceeding $20 billion. Notably, even among those that do survive, many endure significant reductions in physical, emotional and cognitive quality of life. New therapeutic approaches to reduce the high morbidity and mortality of sepsis are needed.

Current management strategies focus on early aggressive fluid resuscitation, blood pressure support with vasopressors, early appropriate antibiotics, and the identification and control of infected sites. Though outcomes have improved with the bundled deployment of these strategies, mortality remains high at 20 - 30%. Despite over a hundred phase 2 and phase 3 clinical trials of pharmacological agents with the potential to improve sepsis outcomes, only antibiotics have demonstrated reproducible benefits.

Despite decades of research, no specific treatment of the dysregulated host response has proven effective. There is strong biologic plausibility to modulate the PCSK9 pathway in sepsis patients. Alirocumab is a PCSK9 inhibitor that has been shown to reduce LDL cholesterol in normal volunteers and in patients with familial hypercholesterolemia.

Patients admitted to a study site hospital with sepsis or septic shock associated with cardiovascular or respiratory failure will be considered for enrollment. Those meeting eligibility criteria and providing consent for study participation will be randomized to receive alirocumab or a placebo, administered once via IV over an approximately 30 ± 10 minute infusion. Participants will be followed for 180 days.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed infection as evidenced by ordering of blood cultures and administration of at least one antimicrobial agent
* Acute respiratory or cardiovascular organ dysfunction attributed to sepsis as evidenced by at least one of the following requirements:

  * Vasopressor Requirement - Continuous infusion of norepinephrine, epinephrine, vasopressin, dopamine, phenylephrine or other vasopressor agents at any dose for greater than 1 hour and required to maintain a mean arterial pressure ≥ 65 mm Hg despite intravenous crystalloid infusion of at least 1000cc
  * Respiratory Support Requirement - Acute hypoxemic respiratory failure defined as persistent hypoxemia requiring (1) intubation and mechanical ventilation, or (2) positive pressure ventilation via tight-fitting face mask or (3) high flow nasal cannula ≥ 45 liters per minute (LPM) flow and fraction of inspired oxygen (FiO2) ≥ 0.40
* Anticipated or confirmed intensive care unit (ICU) admission

Exclusion Criteria:

* Organ dysfunction present > 24 hours at time randomization
* Limitations of care (defined as refusal of cardiovascular and respiratory support described under inclusion criteria) including "do not intubate" (DNI) status
* Development of sepsis while in the hospital ( i.e not present on admission to hospital)
* Chronic hypoxemia requiring supplemental non-invasive oxygen or home mechanical ventilation
* Chronic cardiovascular failure requiring home mechanical hemodynamic support or home chemical hemodynamic support
* Known allergy or known contraindication to alirocumab
* Chronic disease/illness that, in the opinion of the site investigator, have an expected lifespan of < 30 days unrelated to current sepsis diagnosis (e.g, stage IV malignancy, neurodegenerative disease, etc.)
* Requirement of more than 6 liters (L) nasal cannula (NC) if not receiving invasive mechanical ventilation
* Pregnancy
* Prisoner or incarceration
* Current participation in another interventional pharmaceutical research study for sepsis
* Inability or unwillingness of subject or legal surrogate/representative to give written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-23 (Actual)

PRIMARY OUTCOMES:
Bacterial endotoxin level | Hour 120
  Levels of bacterial endotoxin will be compared between study arms.
Lipoteichoic acid level | Hour 120
  Levels of lipoteichoic acid will be compared between study arms.

SECONDARY OUTCOMES:
Number of Vasopressor and Ventilation Free Days (VVFD) | Up to Day 30
  The number of consecutive days free of vasopressors and mechanical ventilation (VVFD) will be compared between study arms. Ventilator and vasopressor free days will only accrue from the last date the participant was free of both ventilator and vasopressor support. Participants who die are scored zero VVFD, and participants who return to ventilator support or vasopressor support will have the VVFD count reset to zero days.
Mortality | Up to Day 30
  The number of participants who die will be compared between study arms.
ICU Mortality | Up to Day 30
  The number of participants who die while in the ICU will be compared between study arms.
Days in ICU | Up to Day 30
  Length of stay in the ICU (measured in days) will be compared between study arms.
Days in Hospital | Up to Day 30
  Length of stay in the hospital (measured in days) will be compared between study arms.
Tumor necrosis factor - alpha (TNF-alpha) Level | Hour 120
  The level of the proinflammatory cytokine TNF will be compared between study arms. Higher levels of TNF are associated with poorer outcomes in patients with sepsis.
Interleukin-1 beta (IL-1 beta) Level | Hour 120
  The level of the proinflammatory cytokine IL-1 will be compared between study arms. Higher levels of IL-1 are associated with poorer outcomes in patients with sepsis.
Interleukin-6 (IL-6) Level | Hour 120
  The level of the proinflammatory cytokine IL-6 will be compared between study arms. Higher levels of IL-6 are associated with poorer outcomes in patients with sepsis.
Interleukin-10 (IL-10) Level | Hour 120
  The level of the proinflammatory cytokine IL-10 will be compared between study arms. Higher levels of IL-10 are associated with poorer outcomes in patients with sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Sevransky, MD, MHS, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data is shared with the funding source (Regeneron) and data will be made available for sharing with other researchers upon request.
Supporting Information: Study Protocol
Time Frame: Individual participant data will be available for sharing one year after publication of the primary manuscript from this study.
Access Criteria: Researchers interested in accessing data from this study should contact the study principal investigator.